CLINICAL TRIAL: NCT00694785
Title: A Study of the Pharmacokinetics, Pharmacodynamics, and Safety of ARC1779 Injection in Patients With Von Willebrand Disease Type 2B
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decided not to go forward with the study.
Sponsor: Archemix Corp. (Industry)
Responsible Party: Margaret Ragni, MD, University of Pittsburgh
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARC1779-010
Record Dates: First submitted 2008-06-06; First posted 2008-06-10 (Estimated); Last update posted 2009-08-21 (Estimated); Status verified 2009-08

CONDITIONS: Von Willebrand Disease
MeSH Terms: conditions — von Willebrand Diseases | interventions — ARC 1779

ARMS (4):
- Group NT3 (Experimental): Patients will receive a total dose of approximately 1.7 mg/kg of ARC1779 over 72 hours to achieve a target plasma concentration of 3 mcg/mL
  Interventions: Drug: ARC1779
- Group T3 (Experimental): Patients will receive a total dose of approximately 1.4 mg/kg of ARC1779 over 72 hours to achieve a target plasma concentration of 3 mcg/mL. The infusion of ARC1779 will be tapered by 50% from 48 hours to 60 hours and again by 50% from 60 hours to 72 hours.
  Interventions: Drug: ARC1779
- Group NT6 (Experimental): Patients will receive a total dose of approximately 3.9 mg/kg of ARC1779 over 72 hours to achieve a target plasma concentration of 6 mcg/mL.
  Interventions: Drug: ARC1779
- Group T6 (Experimental): Patients will receive a total dose of approximately 3.1 mg/kg of ARC1779 over 72 hours to achieve a target plasma concentration of 6 mcg/mL. The infusion of ARC1779 will be tapered by 50% from 48 hours to 60 hours and again by 50% from 60 hours to 72 hours.
  Interventions: Drug: ARC1779

INTERVENTIONS:
Drug: ARC1779 — Initial stepwise infusion of 0.14 mg/kg given over 60 minutes and subsequent continuous infusion of an additional 1.7 mg/kg given over the remaining 72 hours at a rate of 0.0004 mg/kg/min.
  Group "NT3"
  Arms: Group NT3
Drug: ARC1779 — Initial stepwise infusion of 0.14 mg/kg given over 60 minutes and subsequent continuous infusion of an additional 1.3 mg/kg given over the next 72 hours.
  Group "T3"
  Arms: Group T3
Drug: ARC1779 — Initial stepwise infusion of 0.28 mg/kg given over 60 minutes and subsequent continuous infusion of an additional 3.8 mg/kg given over the remaining 72 hours at a rate of 0.0009 mg/kg/min.
  Group "NT6"
  Arms: Group NT6
Drug: ARC1779 — Initial stepwise infusion of 0.28 mg/kg given over 60 minutes and subsequent continuous infusion of an additional 3.0 mg/kg given over the remaining 72 hours.
  Group "T6"
  Arms: Group T6

SUMMARY:
To evaluate the effect of ARC1779, a therapeutic oligonucleotide ("aptamer") in patients with Type2B von Willebrand Disease.

DETAILED DESCRIPTION:
ARC1779 will be investigated in an open-label, uncontrolled study in up to 3 vWD-2B patients. Patients with vWD-2B will be screened for eligibility based primarily upon a single major criterion, i.e., presence of any degree of chronic thrombocytopenia. Eligible patients will be treated by intravenous infusion of ARC1779 for 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients;
* ≥ 16 to ≤ 75 years of age;
* Diagnosis of VWD-2B according to national expert guidelines for the USA [1] and Europe [2] based on medical history and findings from a matrix of laboratory assays which may include: platelet count, concentration of VWF antigen (VWF:Ag), VWF ristocetin cofactor activity (VWF:RCo), Factor VIII (FVIII) activity, ristocetin-induced platelet aggregation (RIPA), platelet function analyzer (PFA-100®) closure time, bleeding time (BT), VWF multimer test, VWF: platelet-binding (VWF:PB) activity, etc.)
* Thrombocytopenia (defined as a platelet count < 100 per nL on at least 2 occasions within the month preceding enrollment;
* Female patients of reproductive age must be enrolled within 1 to 7 days of the cessation of preceding menses;
* Female patients must be non-pregnant and willing to use effective, redundant methods of contraception (i.e., for both self and male partner) throughout the study and for at least 30 days after discontinuation of study drug treatment;
* Male patients must agree to use a medically acceptable contraceptive (abstinence or use of a condom with spermicide) throughout the study and for at least 30 days after discontinuation of study drug treatment;
* All patients must be capable of understanding and complying with the protocol and must have signed the informed consent document.

Exclusion Criteria:

* Patients with a possible co-existing or alternative hematologic diagnosis which can account for the laboratory findings of thrombocytopenia, etc.;
* Any significant medical co-morbidity which would pose an increased risk of bleeding (e.g., recent trauma or surgery, a history of gastrointestinal ulcers, etc.) or thrombosis (e.g., history of recurrent deep vein thrombosis (DVT).

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of ARC1779 Injection on platelet counts in vWD-2B patients who have thrombocytopenia at baseline. | 10 days

SECONDARY OUTCOMES:
To assess the concentration-response relationships among ARC1779 pharmacokinetic (PK) and pharmacodynamic (PD) parameters | 10 days